CLINICAL TRIAL: NCT03217162
Title: Surfactant for Neonate With Acute Respiratory Distress Syndrome (ARDS): A Randomized Controlled Trial
Brief Title: Surfactant for Neonate With Acute Respiratory Distress Syndrome (ARDS)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other)
Responsible Party: Principal Investigator, Ma Juan, Principal Investigator, Daping Hospital and the Research Institute of Surgery of the Third Military Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: surfactant for ARDS
Record Dates: First submitted 2017-07-12; First posted 2017-07-13 (Actual); Last update posted 2022-10-25 (Actual); Status verified 2022-10

CONDITIONS: ARDS; RDS; Surfactant
MeSH Terms: interventions — Respiration, Artificial

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- surfactant combined with mechanical ventilation (Experimental): surfactant is given to the infant with ARDS.
  Interventions: Drug: surfactant combined with mechanical ventilation (MV)
- mechanical ventilation (Active Comparator): mechanical ventilation is given to the infant with ARDS.
  Interventions: Drug: mechanical ventilation (MV)

INTERVENTIONS:
Drug: surfactant combined with mechanical ventilation (MV) — surfactant combined with mechanical ventilation (MV) is given to the infant with ARDS
  Arms: surfactant combined with mechanical ventilation
Drug: mechanical ventilation (MV) — mechanical ventilation (MV) is given to the infant with ARDS
  Arms: mechanical ventilation

SUMMARY:
Acute respiratory distress syndrome (ARDS) in neonates has been defined, the role of surfactant is not clear. This study aimed to determine whether ARDS neonate would benefit from surfactant when oxygenation deteriorated on mechanical ventilation and to identify any potential risk factors related to mortality.

DETAILED DESCRIPTION:
To date, surfactant is not recommended to adult and pediatric ARDS. Meantime, systematic review indicates that surfactant does not demonstrate statistically significant beneficial effects on reducing the mortality and the rate of bronchopulmonary dysplasia(BPD) in term and late preterm infants with meconium aspiration syndrome. Therefore, a reasonable speculation is that preterm infants with ARDS do not benefit from one dose of surfactant. And the speculation can explain why not all preterm infants with respiratory distress can be beneficial from surfactant. In the era of pre-ARDS, the preterm infants fulfilling the definition of ARDS may have been considered as respiratory distress syndrome (ARDS) in the first three days after birth.

According to the diagnostic criteria of neonatal ARDS, a key procedure for diagnosis of neonatal ARDS is to exclude the newborn infants with RDS. But no detailed procedures are available to differentiate RDS from ARDS according the guideline of european RDS and definition of neonatal ARDS.

Therefore, there are two aim in the present study. 1. to proposel a new definition of RDS; 2. to assess the beneficial effects of surfactant on neonatal ARDS.

ELIGIBILITY:
Inclusion Criteria:

1. infant less than 28 days
2. diagnosis of ARDS or RDS or both
3. informed parental consent has been obtained

Exclusion Criteria:

1. major congenital malformations or complex congenital heart disease or chromosomal abnormalities
2. transferred out of the neonatal intensive care unit without treatment
3. upper respiratory tract abnormalities

Ages: 30 Minutes to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2017-08-01 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
death | at 36 weeks' gestational age or before discharge from hospital
  neonates died
bronchopulmonary dysplasia(BPD) | at 36 weeks' gestational age or before discharge from hospital
  neonates were diagnosed with BPD
BPD and/or death | at 36 weeks' gestational age or before discharge from hospital
  neonates were diagnosed with BPD and/or death

SECONDARY OUTCOMES:
Bayley Scales of Infant Development | at 2 months old and 2 years old
  the survival are assessed by Bayley Scales of Infant Development
haemodynamically significant patent ductusarteriosus (hsPDA) | at 36 weeks' gestational age or before discharge from hospital
  neonates were diagnosed with hsPDA
retinopathy of prematurity (ROP)> 2nd stages | at 36 weeks' gestational age or before discharge from hospital
  neonates were diagnosed with ROP> 2nd stages
necrotizing enterocolitis (NEC) ≥ 2nd stages | at 36 weeks' gestational age or before discharge from hospital
  neonates were diagnosed with NEC ≥ 2nd stages
intraventricular hemorrhage(IVH)>2nd grades | at 36 weeks' gestational age or before discharge from hospital
  neonates were diagnosed with IVH >2nd grades

CONTACTS AND LOCATIONS:
Overall Officials: Shi Yuan, PhD,MD, Study Director — Children's Hospital of Chongqing Medical University
Locations (1):
- Department of neonatology, Children's hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided